CLINICAL TRIAL: NCT04071366
Title: A Phase 2 Study of Itacitinib, for the Prevention of Cytokine Release Syndrome Induced by Immune Effector Cell Therapy
Brief Title: A Study of Itacitinib for the Prevention of Cytokine Release Syndrome Induced by Immune Effector Cell Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: INCB 39110-211
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Results first posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-02

CONDITIONS: Cytokine Release Syndrome
Keywords: Cytokine release syndrome; immune effector cell-associated neurotoxicity syndrome; Janus kinase inhibitor; immune effector cell therapy
MeSH Terms: conditions — Cytokine Release Syndrome | interventions — itacitinib; INCB039110; Immunotherapy, Adoptive; axicabtagene ciloleucel

STUDY DESIGN:
Intervention Model Description: Part 1: Singe Group Assignment Part 2: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator
Masking Description: Part 1 is not masked (open label). Part 2 is double blinded (participant, investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Open Label Itacitinib Once Daily (Experimental): During Part 1, all participants receive itacitinib 200mg once daily (open label) for 30 days. The study population will include participants receiving any approved IEC for an approved indication.
  Interventions: Drug: Itacitinib; Drug: Immune effector cell therapy
- Part 2: Double-Blind Itacitinib Twice Daily (Experimental): During Part 2, participants will be randomized to receive itacitinib 200mg or placebo twice daily for 30 days. The study population also includes participants who are receiving Yescarta for relapsed or refractory large B-cell lymphoma or follicular lymphoma.
  Interventions: Drug: Itacitinib; Drug: Placebo; Biological: Yescarta

INTERVENTIONS:
Drug: Itacitinib — Part 1: Itacitinib 200 mg once daily for 30 days. Part 2: Itacitinib 200 mg twice daily for 30 days.
  Other Names: INCB039110
Drug: Immune effector cell therapy — Participants will receive IEC therapy that is approved by the health authority in the country where the study is being conducted for any approved hematologic indication.
  Other Names: CAR-T cell therapy
  Arms: Part 1: Open Label Itacitinib Once Daily
Drug: Placebo — Participants will receive placebo twice daily.
  Arms: Part 2: Double-Blind Itacitinib Twice Daily
Biological: Yescarta — Eligible participants are receiving Yescarta (An infusion of chimeric antigen receptor (CAR)-transduced autologous T cells) for relapsed or refractory larbe B-cell lymphoma or follicular lymphoma intravenously.
  Other Names: axicabtagene ciloleucel KTE-C19
  Arms: Part 2: Double-Blind Itacitinib Twice Daily

SUMMARY:
"The purpose of this study is to assess the safety and efficacy of oral administration of itacitinib for the prevention of cytokine release syndrome (CRS) in male or female participants aged 12 years or older and who are planning to receive an approved immune effector cell (IEC) therapy for hematologic malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Part 1: Eligible to receive any IEC therapy for any approved indication.
* Part 2: Eligible to receive Yescarta for relapsed or refractory large B-cell lymphoma or follicular lymphoma.
* Eastern Cooperative Oncology Group performance status 0 to 1.
* Willingness to avoid pregnancy or fathering children

Exclusion Criteria:

* Evidence of active uncontrolled/untreated infection (viral, bacterial, fungal, opportunistic) of any origin.
* Evidence of active hepatitis B virus or hepatitis C virus infection.
* Known human immunodeficiency virus.
* Active acute or chronic graft-versus-host disease requiring systemic therapy.
* Concurrent use of chronic systemic steroids or immunosuppressant medications.
* Any unresolved toxicity ≥ Grade 2 (except stable Grade 2 peripheral neuropathy or alopecia) from previous anticancer therapy.
* Known history or prior diagnosis of immunologic or inflammatory/autoimmune disease affecting the central nervous system (CNS) and unrelated to their disease under study or previous treatment.
* Clinically significant or uncontrolled cardiac disease.
* Acute lymphoblastic leukemia participants with protocol-defined CNS status are eligible only in the absence of neurologic symptoms suggestive of CNS leukemia.
* Diffuse large B-cell lymphoma participants must have no signs or symptoms of CNS disease or detectable evidence of CNS disease; participants who have been previously treated for CNS disease but have no evidence of disease at screening are eligible.
* Laboratory values at screening outside the protocol-defined ranges.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2020-02-07 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Langmuir, MD, Study Director — Incyte Corporation
Locations (10):
- United States (10):
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Frigault MJ, Maziarz RT, Park JH, Lazaryan A, Shah NN, Svoboda J, Lekakis L, Reshef R, Phillips CL, Burke L, Lei J, Pratta M, Morariu-Zamfir R, DiPersio JF. Itacitinib for the prevention of IEC therapy-associated CRS: results from the 2-part phase 2 INCB 39110-211 study. Blood. 2025 Jul 24;146(4):422-436. doi: 10.1182/blood.2024026586. PMID 40090005
- [Derived] Huarte E, O'Connor RS, Peel MT, Nunez-Cruz S, Leferovich J, Juvekar A, Yang YO, Truong L, Huang T, Naim A, Milone MC, Smith PA. Itacitinib (INCB039110), a JAK1 Inhibitor, Reduces Cytokines Associated with Cytokine Release Syndrome Induced by CAR T-cell Therapy. Clin Cancer Res. 2020 Dec 1;26(23):6299-6309. doi: 10.1158/1078-0432.CCR-20-1739. Epub 2020 Sep 30. PMID 32998963

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1: Itacitinib 200 Milligrams (mg) QD + Kymriah: Participants being treated with Kymriah (Day 0; per prescribing information), an immune effector cell (IEC) therapy for hematologic malignancies, received itacitinib 200 mg once daily (QD) for 30 days (Day -3 to Day 26).
- Part 1: Itacitinib 200 mg QD + Tecartus: Participants being treated with Tecartus (Day 0; per prescribing information), an IEC therapy for hematologic malignancies, received itacitinib 200 mg QD for 30 days (Day -3 to Day 26).
- Part 1: Itacitinib 200 mg QD + Yescarta: Participants being treated with Yescarta (Day 0; per prescribing information), an IEC therapy for hematologic malignancies, received itacitinib 200 mg QD for 30 days (Day -3 to Day 26).
- Part 2: Itacitinib 200 mg BID + Yescarta: Participants being treated with Yescarta (Day 0; per prescribing information) for relapsed or refractory large B-cell lymphoma or follicular lymphoma received itacitinib 200 mg twice daily (BID) for 30 days (Day -3 to Day 26).
- Part 2: Placebo BID + Yescarta: Participants being treated with Yescarta (Day 0; per prescribing information) for relapsed or refractory large B-cell lymphoma or follicular lymphoma BID for 30 days (Day -3 to Day 26).
Period: Part 1: Open-label (29 Days)
Arm/Group | Part 1: Itacitinib 200 Milligrams (mg) QD + Kymriah | Part 1: Itacitinib 200 mg QD + Tecartus | Part 1: Itacitinib 200 mg QD + Yescarta | Part 2: Itacitinib 200 mg BID + Yescarta | Part 2: Placebo BID + Yescarta
Started | 16 | 12 | 35 | 0 | 0
Completed | 11 | 10 | 22 | 0 | 0
Not Completed | 5 | 2 | 13 | 0 | 0
Not completed — Death | 4 | 2 | 8 | 0 | 0
Not completed — Progressive Disease | 0 | 0 | 4 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0 | 0
Period: Part 2: Randomized (29 Days)
Arm/Group | Part 1: Itacitinib 200 Milligrams (mg) QD + Kymriah | Part 1: Itacitinib 200 mg QD + Tecartus | Part 1: Itacitinib 200 mg QD + Yescarta | Part 2: Itacitinib 200 mg BID + Yescarta | Part 2: Placebo BID + Yescarta
Started | 0 | 0 | 0 | 23 | 24
Completed | 0 | 0 | 0 | 17 | 15
Not Completed | 0 | 0 | 0 | 6 | 9
Not completed — Death | 0 | 0 | 0 | 2 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1
Not completed — Progressive Disease | 0 | 0 | 0 | 2 | 4
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0
Not completed — Declined Further Treatment; Entered Hospice | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Itacitinib 200 Milligrams (mg) QD + Kymriah | Part 1: Itacitinib 200 mg QD + Tecartus | Part 1: Itacitinib 200 mg QD + Yescarta | Part 2: Itacitinib 200 mg BID + Yescarta | Part 2: Placebo BID + Yescarta | Total
Number analyzed (Participants) | 16 | 12 | 35 | 23 | 24 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.8 (15.22) | 66.2 (12.08) | 63.5 (10.21) | 63.2 (13.37) | 62.0 (9.93) | 64.18 (11.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 12 | 8 | 7 | 32
  Male | 12 | 11 | 23 | 15 | 17 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 2 | 1 | 0 | 4
  Not Hispanic or Latino | 15 | 10 | 32 | 20 | 23 | 100
  Unknown or Not Reported | 1 | 1 | 1 | 2 | 1 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 13 | 12 | 31 | 21 | 21 | 98
  Black/African-American | 0 | 0 | 2 | 0 | 1 | 3
  Asian | 0 | 0 | 1 | 2 | 1 | 4
  American-Indian/Alaska Native | 1 | 0 | 0 | 0 | 0 | 1
  Captured as "Other" in Database | 2 | 0 | 1 | 0 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Developed ≥Grade 2 Cytokine Release Syndrome (CRS) by Day 14 After Immune Effector Cell (IEC) Therapy, Assessed by Using American Society for Blood and Marrow Transplantation (ASBMT) CRS Consensus Grading
Description: The ASBMT CRS Consensus Grading Criteria was used to assess the severity of CRS. Grade 2 CRS: temperature ≥38°C not attributable to any other cause, defined as fever; hypotension not requiring vasopressors, and/or; hypoxia requiring low-flow nasal cannula (oxygen delivered at ≤6 liters/minute) or blow-by. Grade 3 CRS: fever; hypotension requiring one vasopressor with or without vasopressin, and/or; hypoxyia requiring high-flow nasal cannula (oxygen delivered at >6 liters/minute), facemask, nonrebreather mask, or Venturi mask. Grade 4 CRS: fever; hypotension requiring multiple vasopressors (excluding vasopressin), and/or; hypoxia requiring positive pressure (e.g., continuous positive airway pressure [CPAP], bilevel intermittent positive air pressure [BiPAP], intubation, mechanical ventilation).
Time Frame: up to Day 14 of Parts 1 and 2
Population: Efficacy Evaluable Analysis Set (EAS): all participants who received at least 1 dose of study drug and received IEC therapy. The exact 95% confidence interval (2-sided) was calculated using the Clopper-Pearson method.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: Itacitinib 200 Milligrams (mg) QD + Kymriah | Part 1: Itacitinib 200 mg QD + Tecartus | Part 1: Itacitinib 200 mg QD + Yescarta | Part 2: Itacitinib 200 mg BID + Yescarta | Part 2: Placebo BID + Yescarta
Number analyzed (Participants) | 16 | 12 | 35 | 23 | 23
percentage of participants | 12.5 [1.6 to 38.3] | 41.7 [15.2 to 72.3] | 20.0 [8.4 to 36.9] | 17.4 [5.0 to 38.8] | 56.5 [34.5 to 76.8]
Statistical Analysis 1: Comparison: Part 2: Itacitinib 200 mg BID + Yescarta vs Part 2: Placebo BID + Yescarta; Test type: Superiority; p = 0.0030, One-sided Z-test; Difference in CRS rate = -0.39, 95% CI 2-sided [-0.6463 to -0.1363]
Statistical Analysis 2: Comparison: Part 1: Itacitinib 200 mg QD + Yescarta vs Part 2: Placebo BID + Yescarta; Test type: Other; Difference in CRS rate = -0.37, 95% CI 2-sided [-0.6073 to -0.1231]
Statistical Analysis 3: Comparison: Part 1: Itacitinib 200 mg QD + Yescarta vs Part 2: Itacitinib 200 mg BID + Yescarta; Test type: Other; Difference in CRS rate = 0.03, 95% CI 2-sided [-0.1778 to 0.2299]

2. Secondary Outcome: Percentage of Participants With Immune Effector Cell-associated Neurotoxicity Syndrome (ICANS) by Day 28 After IEC Therapy, Assessed by Using the ICANS Consensus Grading
Description: Participants were monitored for signs and symptoms of ICANS, if symptoms developed at any point after IEC. ICANS Consensus Grading Criteria were used to assess 5 domains of neurotoxicity: orientation (orient to year, month, city, and hospital), naming (naming 3 objects), following commands (follow commands such as: show me 2 fingers or close your eyes and stick out your tongue), writing (ability to write a standard sentence), and attention (count backwards from 100 by 10). Each domain is associated with a certain number of points, which are summed to generate a total score. Score 10: no impairment; score 7-9: Grade 1 ICANS; score 3-6: Grade 2 ICANS; score 0-2: Grade 3 ICANS.
Time Frame: up to Day 28 of Parts 1 and 2
Population: EAS. The exact 95% confidence interval (2-sided) was calculated using the Clopper-Pearson method.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: Itacitinib 200 Milligrams (mg) QD + Kymriah | Part 1: Itacitinib 200 mg QD + Tecartus | Part 1: Itacitinib 200 mg QD + Yescarta | Part 2: Itacitinib 200 mg BID + Yescarta | Part 2: Placebo BID + Yescarta
Number analyzed (Participants) | 16 | 12 | 35 | 23 | 23
percentage of participants | 31.3 [11.0 to 58.7] | 41.7 [15.2 to 72.3] | 45.7 [28.8 to 63.4] | 13.0 [2.8 to 33.6] | 34.8 [16.4 to 57.3]

3. Secondary Outcome: Time to Onset of ICANS Using the ICANS Consensus Grading, Regardless of CRS, by Day 28 After IEC Therapy
Description: as for outcome 2
Time Frame: up to Day 28 of Parts 1 and 2
Population: EAS. Only participants with ICANS onset by Day 28 were analyzed.
Measure: Median (Full Range); unit: days
Arm/Group | Part 1: Itacitinib 200 Milligrams (mg) QD + Kymriah | Part 1: Itacitinib 200 mg QD + Tecartus | Part 1: Itacitinib 200 mg QD + Yescarta | Part 2: Itacitinib 200 mg BID + Yescarta | Part 2: Placebo BID + Yescarta
Number analyzed (Participants) | 5 | 5 | 16 | 3 | 8
days | 4.0 [0 to 11] | 4.0 [0 to 6] | 5.0 [1 to 9] | 5.0 [4 to 9] | 6.5 [2 to 11]

4. Secondary Outcome: Duration of ICANS Occurring by Day 28 After IEC Therapy Using the ICANS Consensus Grading, Regardless of CRS
Description: Participants were monitored for signs and symptoms of ICANS, if symptoms developed at any point after IEC. ICANS Consensus Grading Criteria were used to assess 5 domains of neurotoxicity: orientation (orient to year, month, city, and hospital), naming (naming 3 objects), following commands (follow commands such as: show me 2 fingers or close your eyes and stick out your tongue), writing (ability to write a standard sentence), and attention (count backwards from 100 by 10). Each domain is associated with a certain number of points, which are summed to generate a total score. Score 10: no impairment; score 7-9: Grade 1 ICANS; score 3-6: Grade 2 ICANS; score 0-2: Grade 3 ICANS. Duration of ICANS occurring by Day 28 corresponds to the sum of days with non-zero grade ICANS by Day 28.
Time Frame: up to Day 28 of Parts 1 and 2
Population: EAS. Only participants with ICANS onset by Day 28 were analyzed.
Measure: Median (Full Range); unit: days
Arm/Group | Part 1: Itacitinib 200 Milligrams (mg) QD + Kymriah | Part 1: Itacitinib 200 mg QD + Tecartus | Part 1: Itacitinib 200 mg QD + Yescarta | Part 2: Itacitinib 200 mg BID + Yescarta | Part 2: Placebo BID + Yescarta
Number analyzed (Participants) | 5 | 5 | 16 | 3 | 8
days | 3.0 [1 to 4] | 5.0 [1 to 17] | 1.5 [1 to 16] | 2.0 [2 to 11] | 3.5 [2 to 13]

5. Secondary Outcome: Time to Onset of All Grades of CRS by Day 28 After IEC Therapy, Assessed by Using ASBMT CRS Consensus Grading
Description: The ASBMT CRS Consensus Grading Criteria was used to assess the severity of CRS. Grade 1: fever; either no hypotention and/or no hypoxia. Grade 2 CRS: fever; hypotension not requiring vasopressors, and/or; hypoxia requiring low-flow nasal cannula (oxygen delivered at ≤6 liters/minute) or blow-by. Grade 3 CRS: fever; hypotension requiring one vasopressor with or without vasopressinc, and/or; hypoxyia requiring high-flow nasal cannula (oxygen delivered at >6 liters/minute), facemask, nonrebreather mask, or Venturi mask. Grade 4 CRS: fever; hypotension requiring multiple vasopressors (excluding vasopressin), and/or; hypoxia requiring positive pressure (e.g., CPAP, BiPAP, intubation, mechanical ventilation).
Time Frame: up to Day 28 of Parts 1 and 2
Population: EAS. Only participants with CRS onset by Day 28 were analyzed.
Measure: Median (Full Range); unit: days
Arm/Group | Part 1: Itacitinib 200 Milligrams (mg) QD + Kymriah | Part 1: Itacitinib 200 mg QD + Tecartus | Part 1: Itacitinib 200 mg QD + Yescarta | Part 2: Itacitinib 200 mg BID + Yescarta | Part 2: Placebo BID + Yescarta
Number analyzed (Participants) | 14 | 10 | 30 | 15 | 20
days | 2.0 [1 to 6] | 2.5 [0 to 7] | 1.0 [1 to 8] | 2.0 [0 to 8] | 3.0 [0 to 9]

6. Secondary Outcome: Duration of All Grades of CRS Occurring by Day 28 After IEC Therapy, Assessed by Using ASBMT CRS Consensus Grading
Description: as for outcome 5
Time Frame: up to Day 56 of Parts 1 and 2
Population: EAS. Only participants with CRS onset by Day 28 were analyzed.
Measure: Median (Full Range); unit: days
Arm/Group | Part 1: Itacitinib 200 Milligrams (mg) QD + Kymriah | Part 1: Itacitinib 200 mg QD + Tecartus | Part 1: Itacitinib 200 mg QD + Yescarta | Part 2: Itacitinib 200 mg BID + Yescarta | Part 2: Placebo BID + Yescarta
Number analyzed (Participants) | 14 | 10 | 30 | 15 | 20
days | 5.0 [2 to 11] | 4.0 [2 to 11] | 5.0 [1 to 11] | 5.0 [3 to 12] | 4.0 [1 to 8]

7. Secondary Outcome: Percentage of Participants With Any Grade of CRS at 48 Hours After IEC Therapy, Assessed by Using ASBMT CRS Consensus Grading
Description: as for outcome 5
Time Frame: up to Day 2 of Parts 1 and 2
Population: EAS. The exact 95% confidence interval (2-sided) was calculated using the Clopper-Pearson method.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: Itacitinib 200 Milligrams (mg) QD + Kymriah | Part 1: Itacitinib 200 mg QD + Tecartus | Part 1: Itacitinib 200 mg QD + Yescarta | Part 2: Itacitinib 200 mg BID + Yescarta | Part 2: Placebo BID + Yescarta
Number analyzed (Participants) | 16 | 12 | 35 | 23 | 23
percentage of participants | 37.5 [15.2 to 64.6] | 33.3 [9.9 to 65.1] | 48.6 [31.4 to 66.0] | 26.1 [10.2 to 48.4] | 30.4 [13.2 to 52.9]

8. Secondary Outcome: Percentage of Participants With ≥Grade 2 CRS by Day 28 After First IEC Therapy, Assessed by Using ASBMT CRS Consensus Grading
Description: as for outcome 5
Time Frame: up to Day 28 of Parts 1 and 2
Population: EAS. The exact 95% confidence interval (2-sided) was calculated using the Clopper-Pearson method.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: Itacitinib 200 Milligrams (mg) QD + Kymriah | Part 1: Itacitinib 200 mg QD + Tecartus | Part 1: Itacitinib 200 mg QD + Yescarta | Part 2: Itacitinib 200 mg BID + Yescarta | Part 2: Placebo BID + Yescarta
Number analyzed (Participants) | 16 | 12 | 35 | 23 | 23
percentage of participants | 12.5 [1.6 to 38.3] | 41.7 [15.2 to 72.3] | 20.0 [8.4 to 36.9] | 21.7 [7.5 to 43.7] | 56.5 [34.5 to 76.8]

9. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE) Except CRS and ICANS
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study treatment. For purposes of analysis, all AEs were considered TEAEs unless the AE could unequivocally be defined as not treatment emergent.
Time Frame: from at Day -3 through the duration of safety follow-up (up to Day 56) for Parts 1 and 2
Population: Safety Evaluable Set: all enrolled participants who received at least 1 dose of study drug
Measure: Number; unit: participants
Arm/Group | Part 1: Itacitinib 200 Milligrams (mg) QD + Kymriah | Part 1: Itacitinib 200 mg QD + Tecartus | Part 1: Itacitinib 200 mg QD + Yescarta | Part 2: Itacitinib 200 mg BID + Yescarta | Part 2: Placebo BID + Yescarta
Number analyzed (Participants) | 16 | 12 | 35 | 23 | 24
participants | 16 | 12 | 35 | 22 | 24

10. Secondary Outcome: Percentage of Participants With Any ≥Grade 3 Cytopenias Ongoing at Day 28
Description: Cytopenia is characterized by low levels of white blood cells, red blood cells, or platelets. Analysis used laboratory counts at Day 28.
Time Frame: Day 28 of Parts 1 and 2
Population: EAS. Only participants with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: Itacitinib 200 Milligrams (mg) QD + Kymriah | Part 1: Itacitinib 200 mg QD + Tecartus | Part 1: Itacitinib 200 mg QD + Yescarta | Part 2: Itacitinib 200 mg BID + Yescarta | Part 2: Placebo BID + Yescarta
Number analyzed (Participants) | 16 | 12 | 35 | 23 | 23
percentage of participants
  Neutrophils: number analyzed (Participants) | 16 | 12 | 35 | 22 | 23
  Neutrophils | 8.3 | 22.2 | 26.6 | 31.8 | 13.6
  Hemoglobin: number analyzed (Participants) | 16 | 12 | 35 | 22 | 23
  Hemoglobin | 0.0 | 20.0 | 16.7 | 9.1 | 4.5
  Platelets: number analyzed (Participants) | 16 | 12 | 35 | 22 | 23
  Platelets | 25.0 | 50.0 | 26.7 | 36.4 | 18.2

11. Other Pre Specified Outcome: Number of Hospital Admissions for Participants With CRS and/or ICANS by the End of the Study
Description: The number of hospital admissions was assessed through study completion.
Time Frame: up to Day 180 of Parts 1 and 2
Population: Data have not been reported, as the outcome measure is exploratory.
Arm/Group | Part 1: Itacitinib 200 Milligrams (mg) QD + Kymriah | Part 1: Itacitinib 200 mg QD + Tecartus | Part 1: Itacitinib 200 mg QD + Yescarta | Part 2: Itacitinib 200 mg BID + Yescarta | Part 2: Placebo BID + Yescarta
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

12. Other Pre Specified Outcome: Duration of Hospital Stay for Participants With CRS and/or ICANS by End of Study
Description: The duration of hospital stays was assessed through study completion.
Time Frame: up to Day 180 of Parts 1 and 2
Population: Data have not been reported as the outcome measure is exploratory.
Arm/Group | Part 1: Itacitinib 200 Milligrams (mg) QD + Kymriah | Part 1: Itacitinib 200 mg QD + Tecartus | Part 1: Itacitinib 200 mg QD + Yescarta | Part 2: Itacitinib 200 mg BID + Yescarta | Part 2: Placebo BID + Yescarta
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Percentage of Participants Who Were Treated With Tocilizumab for CRS
Description: Tocilizumab and/or corticosteroids for CRS Grade 1 was not allowed per the protocol. However, tocilizumab may have been given as rescue medication for CRS Grade 1 if no improvement was observed within 72 hours from onset, and the participant's medical condition required intervention per investigator judgment.
Time Frame: up to Day 56 of Parts 1 and 2
Population: EAS
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: Itacitinib 200 Milligrams (mg) QD + Kymriah | Part 1: Itacitinib 200 mg QD + Tecartus | Part 1: Itacitinib 200 mg QD + Yescarta | Part 2: Itacitinib 200 mg BID + Yescarta | Part 2: Placebo BID + Yescarta
Number analyzed (Participants) | 16 | 12 | 35 | 23 | 23
percentage of participants | 18.8 | 41.7 | 20.0 | 17.4 | 65.2

14. Secondary Outcome: Percentage of Participants Requiring More Than 1 Dose of Dexamethasone (or Equivalent) for ICANS
Description: Dexamethasone use as rescue medication for ICANS was assessed.
Time Frame: up to Day 30 of Parts 1 and 2
Population: EAS
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: Itacitinib 200 Milligrams (mg) QD + Kymriah | Part 1: Itacitinib 200 mg QD + Tecartus | Part 1: Itacitinib 200 mg QD + Yescarta | Part 2: Itacitinib 200 mg BID + Yescarta | Part 2: Placebo BID + Yescarta
Number analyzed (Participants) | 16 | 12 | 35 | 23 | 23
percentage of participants | 12.5 | 25.0 | 22.9 | 4.3 | 30.4

ADVERSE EVENTS:
Time Frame: TEAEs collected from Day -3 through the duration of safety follow-up (up to Day 56) for Parts 1 and 2 have been reported. Deaths occurring up to the end of the study (Day 180) or until early study withdrawal have been reported.
Description: Treatment-emergent adverse events (TEAES), defined as any AEs unless the AEs could unequivocally be defined as not treatment emergent, have been reported for members of the Safety Evaluable Set (all enrolled participants who received at least 1 dose of study drug).
Groups:
- Part 1: Itacitinib 200 mg + Any IEC: Participants being treated with Kymriah, Yescarta, and Tecartus (Day 0; per prescribing information), IEC therapies for hematologic malignancies, received itacitinib 200 mg once daily for 30 days (Day -3 to Day 26).
Arm/Group | Part 1: Itacitinib 200 Milligrams (mg) QD + Kymriah | Part 1: Itacitinib 200 mg QD + Tecartus | Part 1: Itacitinib 200 mg QD + Yescarta | Part 1: Itacitinib 200 mg + Any IEC | Part 2: Itacitinib 200 mg BID + Yescarta | Part 2: Placebo BID + Yescarta
All-Cause Mortality (participants affected / at risk) | 4/16 | 2/12 | 9/35 | 15/63 | 2/23 | 2/24
Serious Adverse Events (participants affected / at risk) | 2/16 | 1/12 | 9/35 | 12/63 | 3/23 | 6/24
Other Adverse Events (participants affected / at risk) | 16/16 | 12/12 | 35/35 | 63/63 | 22/23 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Itacitinib 200 Milligrams (mg) QD + Kymriah (N=16) | Part 1: Itacitinib 200 mg QD + Tecartus (N=12) | Part 1: Itacitinib 200 mg QD + Yescarta (N=35) | Part 1: Itacitinib 200 mg + Any IEC (N=63) | Part 2: Itacitinib 200 mg BID + Yescarta (N=23) | Part 2: Placebo BID + Yescarta (N=24)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fusarium infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Immune effector cell-associated neurotoxicity syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neurotoxicity (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pneumonia necrotising (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Sinusitis fungal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VIth nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Itacitinib 200 Milligrams (mg) QD + Kymriah (N=16) | Part 1: Itacitinib 200 mg QD + Tecartus (N=12) | Part 1: Itacitinib 200 mg QD + Yescarta (N=35) | Part 1: Itacitinib 200 mg + Any IEC (N=63) | Part 2: Itacitinib 200 mg BID + Yescarta (N=23) | Part 2: Placebo BID + Yescarta (N=24)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 5 (5) | 6 (6) | 1 (2) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 1 (2) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Affect lability (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 1 (2) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 5 (5)
Amylase increased (Investigations) | 0 (0) | 2 (3) | 1 (1) | 3 (4) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 7 (9) | 5 (8) | 9 (14) | 21 (31) | 5 (9) | 6 (7)
Anal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1) | 2 (2) | 5 (5) | 1 (1) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 3 (3) | 6 (6) | 1 (1) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 2 (3) | 4 (5) | 3 (3) | 3 (3)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 3 (3) | 8 (8) | 2 (2) | 4 (5)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 2 (2) | 2 (2) | 5 (5) | 1 (1) | 3 (3)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Blood fibrinogen decreased (Investigations) | 0 (0) | 1 (1) | 1 (2) | 2 (3) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 3 (5) | 1 (1) | 5 (7) | 0 (0) | 2 (2)
C-reactive protein increased (Investigations) | 0 (0) | 3 (5) | 1 (1) | 4 (6) | 0 (0) | 0 (0)
Catheter site haemorrhage (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site related reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 6 (8) | 4 (5) | 8 (8) | 18 (21) | 9 (12) | 6 (6)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 2 (2) | 4 (4) | 7 (7) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 6 (9) | 4 (4) | 7 (7) | 17 (20) | 6 (7) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 4 (4) | 9 (9) | 1 (1) | 5 (5)
Cytomegalovirus viraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 8 (11) | 4 (4) | 4 (4) | 16 (19) | 5 (5) | 7 (7)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 4 (4) | 1 (1)
Delirium febrile (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 8 (9) | 4 (4) | 6 (6) | 18 (19) | 5 (8) | 7 (7)
Disorganised speech (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 2 (2) | 6 (7) | 11 (12) | 4 (6) | 5 (6)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 2 (3) | 2 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 6 (6) | 7 (7) | 2 (3) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Electrocardiogram QT prolonged (Investigations) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Facial pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 4 (4) | 5 (5) | 1 (1) | 0 (0)
Fatigue (General disorders) | 8 (9) | 6 (7) | 18 (18) | 32 (34) | 7 (8) | 10 (10)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (3) | 1 (1) | 2 (2) | 5 (6) | 4 (6) | 3 (3)
Fluid intake reduced (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 7 (8) | 7 (8) | 12 (14) | 26 (30) | 6 (8) | 8 (8)
Hyperaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 4 (7)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 4 (6) | 1 (1) | 0 (0) | 5 (7) | 1 (1) | 3 (5)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 2 (5) | 5 (9) | 1 (1) | 4 (5)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (3) | 2 (2) | 2 (2) | 6 (7) | 2 (3) | 5 (6)
Hypogammaglobulinaemia (Immune system disorders) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (5) | 3 (6) | 8 (11) | 14 (22) | 4 (4) | 4 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (7) | 3 (3) | 7 (11) | 3 (6) | 2 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 3 (4) | 7 (8) | 4 (8) | 5 (5)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 3 (6) | 2 (5) | 11 (12) | 16 (23) | 1 (3) | 4 (4)
Hypotension (Vascular disorders) | 3 (3) | 4 (4) | 14 (18) | 21 (25) | 8 (12) | 9 (11)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 5 (5) | 7 (7) | 3 (3) | 5 (5)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 6 (7) | 5 (5) | 14 (15) | 2 (2) | 4 (4)
Klebsiella infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 3 (4) | 1 (1) | 4 (5) | 0 (0) | 1 (2)
Lymphocyte count decreased (Investigations) | 2 (4) | 3 (4) | 6 (9) | 11 (17) | 8 (13) | 7 (12)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2) | 2 (3) | 0 (0) | 4 (5) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mental impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 1 (1) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 4 (4) | 8 (8) | 0 (0) | 1 (1)
Myoclonus (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 5 (5) | 5 (7) | 15 (21) | 25 (33) | 6 (9) | 10 (10)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neurotoxicity (Nervous system disorders) | 1 (1) | 1 (1) | 2 (4) | 4 (6) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 3 (6) | 3 (5) | 3 (3) | 9 (14) | 2 (2) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (3) | 2 (2) | 8 (14) | 12 (19) | 9 (19) | 7 (11)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Oedema (General disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 5 (5) | 0 (0) | 3 (3) | 8 (8) | 0 (0) | 2 (2)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 1 (2) | 3 (3) | 5 (6) | 2 (2) | 1 (1)
Pain (General disorders) | 3 (3) | 0 (0) | 2 (2) | 5 (5) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
Penile ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 4 (6) | 2 (3) | 6 (10) | 12 (19) | 4 (5) | 4 (8)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Polyomavirus viraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 8 (13) | 8 (12) | 22 (25) | 38 (50) | 10 (13) | 12 (14)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 2 (2)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sensitive skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Serum ferritin increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 5 (6) | 7 (8) | 3 (3) | 3 (4)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (3) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 1 (2) | 5 (5) | 8 (9) | 2 (2) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (3) | 3 (3) | 2 (3) | 7 (9) | 2 (3) | 0 (0)
Tremor (Nervous system disorders) | 2 (2) | 0 (0) | 5 (5) | 7 (7) | 3 (3) | 7 (8)
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 0 (0) | 2 (2) | 4 (4) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Vision blurred (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (5) | 2 (2) | 3 (4) | 7 (11) | 3 (4) | 4 (4)
Weight decreased (Investigations) | 3 (5) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 2 (3) | 6 (10) | 8 (13) | 6 (12) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2022-12-08): https://cdn.clinicaltrials.gov/large-docs/66/NCT04071366/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-08): https://cdn.clinicaltrials.gov/large-docs/66/NCT04071366/SAP_001.pdf